CLINICAL TRIAL: NCT02107794
Title: Shared Decision Making in Graves Disease - Graves Disease (GD) Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 12-007708
Record Dates: First submitted 2014-03-24; First posted 2014-04-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Graves' Disease; Thyroid Disease; Hyperthyroidism
Keywords: Grave's; Disease; Thyroid; Hyperthyroidism; Thyroidectomy; Radioactive; Iodine; Antithyroid; Shared; Decision; Making; Aid; Evidence; Based; Endocrinology; Mayo; Clinic
MeSH Terms: conditions — Graves Disease; Thyroid Diseases; Hyperthyroidism; Disease; Helping Behavior | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Active Comparator): Observation of clinical encounter using the decision aid, via video, audio or written notes.
  Interventions: Other: Decision Aid
- Usual Care (No Intervention): Observations in clinical encounters, either video, audio, or observational notes.

INTERVENTIONS:
Other: Decision Aid — Paper based decision aid will be utilized to facilitate treatment option conversation between clinician and patient.
  Other Names: DA
  Arms: Decision Aid

SUMMARY:
The investigators' decision aid for patients with GD, GD Choice, will be the result of a user-centered participatory action research involving) synthesis of the best available evidence from the literature and real-world registry experience, ii) input and involvement of patients, clinicians and other stakeholders, iii) direct observation of encounters and iv) extensive field-testing. The goal is to create a decision aid that will be rigorously evidence-based, clear and complete, able to be used by clinicians with minimal training time, while satisfying extant standards for rigorous high-quality shared decision making tools.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Diagnosis of Graves Disease
* Appointment with endocrinologist to discuss treatment options for Graves Disease

Exclusion Criteria:

* Major barriers to participate in shared decision making or to providing informed consent (i.e. dementia, severe hearing or visual impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Decisional Quality (Knowledge, Decisional Conflict, Satisfaction) of 100 participants | up to 2 weeks post-visit
  Outcome measure to be assessed through post-visit surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Montori, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Brito JP, Castaneda-Guarderas A, Gionfriddo MR, Ospina NS, Maraka S, Dean DS, Castro MR, Fatourechi V, Gharib H, Stan MN, Branda ME, Bahn RS, Montori VM. Development and Pilot Testing of an Encounter Tool for Shared Decision Making About the Treatment of Graves' Disease. Thyroid. 2015 Nov;25(11):1191-8. doi: 10.1089/thy.2015.0277. Epub 2015 Oct 15. PMID 26413979